CLINICAL TRIAL: NCT02345694
Title: Non-automatic Control of Gait and Posture in Obstructive Sleep Apnea Syndrome : a Randomised Controlled Trial of Continuous Positive Airway Pressure Effectiveness (CIH - Gait)
Brief Title: Non-automatic Control of Gait and Posture in Obstructive Sleep Apnea Syndrome (CIH-Gait)
Acronym: CIH-Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Agence Régionale de Santé Rhône-Alpes (Other)
Responsible Party: Principal Investigator, AdministrateurDRC, Directeur de la recherche clinique, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2014-A01523-44
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; Gait; Posture; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Effective CPAP (Experimental): Continuous Positive Airway Pressure (RESMED S9™ Series), all the nights, during 8 weeks.
  Interventions: Device: Effective CPAP
- Sub-therapeutic CPAP (Sham Comparator): Sub-therapeutic Continuous Positive Airway Pressure (RESMED S9™ Sham-Continuous Positive Airway Pressure System), validated placebo of Continuous Positive Airway Pressure, all the nights, during 8 weeks.
  Interventions: Device: Sub-therapeutic CPAP

INTERVENTIONS:
Device: Effective CPAP — Effective Continuous Positive Airway Pressure auto-regulated, worn all night long during 8 weeks
  Other Names: Continuous positive airway pressure (RESMED S9™ Series)
  Arms: Effective CPAP
Device: Sub-therapeutic CPAP — Sub-therapeutic Continuous Positive Airway Pressure (Sham-CPAP) worn all night long during 8 weeks
  Other Names: Sham-CPAP (RESMED S9™ Sham-CPAP System)
  Arms: Sub-therapeutic CPAP

SUMMARY:
The purpose of this randomised controlled study is to determine the impact of continuous positive airway pressure (CPAP) versus sub-therapeutic CPAP (placebo) on the control of gait upon severe sleep apnea patients, based on stride time variability.

DETAILED DESCRIPTION:
As severe sleep apnea patients exhibit gait abnormalities, this is the first randomised controlled trial to our knowledge to assess the impact of CPAP upon gait and postural control in severe sleep apnea patients. Based on a dual-task paradigm, posture and gait analysis will be perform before and after 8 week of intervention.

Beside gait parameters, the cerebral metabolism will be assessed using a Near Infrared Spectroscopy (fNIRS) device during normal walking and during walking while dual-tasking, using a visual and a verbal task.

ELIGIBILITY:
Inclusion Criteria:

* Normally weighted or over-weighted patients (BMI < 30 kilograms/m²)
* Newly diagnosed Obstructive Sleep Apnea Syndrome (OSAS) (i.e. no previous treatment)
* Severe OSAS as defined by the American Academy of Sleep Medicine (AHI ≥ 30)
* To speak and understand french
* To be affiliated to social welfare

Exclusion Criteria:

* Age criteria : <18 year old and >70 year old
* Obesity (BMI ≥ 30 kilograms/m²)
* Pathological conditions thought to be responsible of gait unsteadiness and postural sway or requiring an walking device : nervous system disease (Parkinson disease, chronic stroke), cerebellum syndrome, vestibular syndrome, orthopaedic and rheumatic diseases,
* Lower limb sensitivity impairment,
* Cognitive disorder (Folstein test score < 24),
* Ophthalmology disorder : uncorrected refractive disorder, disturbance of color vision,
* Psychotropic treatment intake,
* Alcoholism,
* Member of an at-risk occupation (car, bus, truck drivers...) mandating effective continuous positive airway pressure introduction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of stride time coefficient of variation at 8 weeks | Baseline and 8 weeks
  The stride time will be recorded during an overground walking test, under single (walking alone) and dual-task (walking while performing a cognitive task) condition. The cognitive task used in our protocol is an electronic Stroop test, displayed on a screen at the end of the 10 meters walkway. The coefficient of variation allows us to estimate stride time variability, known to be the reflect of gait control efficiency when it exhibits low values.

SECONDARY OUTCOMES:
Change from baseline of single support time and percentage at 8 weeks | Baseline and 8 weeks
  To assess gait stability, mean single support time will be assess under single (walking alone) and dual task condition (walking while performing a cognitive task) and its coefficient of variation calculate.
Change from baseline of double support time and percentage at 8 weeks | Baseline and 8 weeks
  To assess gait stability, mean double support time will be assess and its coefficient of variation calculate.
Change from baseline of gait speed at 8 weeks | Baseline and 8 weeks
Change from baseline of step length at 8 weeks | Baseline and 8 weeks
Change from baseline of step width at 8 weeks | Baseline and 8 weeks
Change from baseline of the center-of-pressure area at 8 weeks | Baseline and 8 weeks
  Studying gait implies posture assessment as the link between gait stability and an efficient postural control is tenuous.
Change from baseline of the center-of-pressure length at 8 weeks | Baseline and 8 weeks
  Combined with center-of-pressure (CoP) area, the length (path of CoP) of CoP permits efficient measurement of CoP spatial variability.
Change from baseline of the center-of-pressure mean speed at 8 weeks | Baseline and 8 weeks
  The mean speed represents a good index of the amount of neuromuscular activity required to regulate postural control.
Change from baseline of oxy-haemoglobin concentration of bilateral prefrontal cortices at 8 weeks | Baseline and 8 weeks
  The oxyhaemoglobin concentration will be recorded during an treadmill walking test, under single (walking alone) and dual-task (walking while performing a cognitive task) condition. The cognitive task used in our protocol is an electronic Stroop test, displayed on a screen placed in front of the patient.
  We use a fNIRS (Near Infrared Spectroscopy) device, disposed bilaterally opposite to prefrontal cortices to assess the change of oxyhemoglobin concentration over different motor and cognitive tasks.
Change from baseline of deoxy-haemoglobin concentration of bilateral prefrontal cortices at 8 weeks | Baseline and 8 weeks
  The deoxyhemoglobin concentration will be recorded as oxyhaemoglobin concentration.
Change from baseline of total haemoglobin concentration of bilateral prefrontal cortices at 8 weeks | Baseline and 8 weeks
  The total haemoglobin concentration will be recorded as oxyhaemoglobin concentration.

OTHER OUTCOMES:
Change from baseline in Dual Task Cost (DTC) at 8 weeks | Baseline and 8 weeks
  Dual Task Cost = [(Dual Task % correct - Single Task % correct) x 100 / Single Task % correct]
Continuous Positive Airway Pressure Observance at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernard WUYAM, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Institut de rééducation, Hôpital Sud, CHU de GRENOBLE, Échirolles, Isère, France

REFERENCES:
- [Background] Allali G, Perrig S, Cleusix M, Herrmann FR, Adler D, Gex G, Armand S, Janssens JP, Pepin JL, Assal F. Gait abnormalities in obstructive sleep apnea and impact of continuous positive airway pressure. Respir Physiol Neurobiol. 2014 Sep 15;201:31-3. doi: 10.1016/j.resp.2014.06.012. Epub 2014 Jul 4. PMID 24999279
- [Background] Celle S, Annweiler C, Camicioli R, Barthelemy JC, Roche F, Beauchet O. Sleep-related breathing disorders and gait variability: a cross-sectional preliminary study. BMC Pulm Med. 2014 Aug 23;14:140. doi: 10.1186/1471-2466-14-140. PMID 25150985
- [Derived] Baillieul S, Wuyam B, Perennou D, Tamisier R, Bailly S, Benmerad M, Piscicelli C, Le Roux-Mallouf T, Verges S, Pepin JL. A randomized sham-controlled trial on the effect of continuous positive airway pressure treatment on gait control in severe obstructive sleep apnea patients. Sci Rep. 2021 Apr 29;11(1):9329. doi: 10.1038/s41598-021-88642-5. PMID 33927278